CLINICAL TRIAL: NCT03908294
Title: Examination of Changes of Parameters of Glucose Metabolism and Liver Fibrosis Stadium by Acoustic Radiation Force Impulse-Imaging and Transient Elastography in Patients With Chronic Hepatitis C Under Antiviral Treatment
Brief Title: Change of Glucose Metabolism and Fibrosis Markers in Patients With Hepatitis C Under Treatment With Antiviral Agents
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, Prof., Johann Wolfgang Goethe University Hospital
Other Study IDs: JWGUHMED1-012
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Glucose Metabolism Disorders; Liver Fibrosis; Hepatitis C
MeSH Terms: conditions — Glucose Metabolism Disorders; Liver Cirrhosis; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hepatitis C under antiviral treatment with DAA: Patients with chronic hepatitis C infection and planned DAA treatment are enrolled prospectively. Parameters of glucose metabolism and liver fibrosis are measured at baseline, during therapy and up to one year after end of treatment.
  Interventions: Diagnostic Test: Lab tests, non-invasive fibrosis (Fibroscan/ARFI)

INTERVENTIONS:
Diagnostic Test: Lab tests, non-invasive fibrosis (Fibroscan/ARFI) — Patient characteristics, lab values reflecting glucose metabolism and non-invasive fibrosis tests are documented at baseline, during therapy and up to one year after end of treatment.

SUMMARY:
Chronic hepatitis C infection is associated with changes of glucose metabolism end increased frequency of impaired glucose tolerance. This might be a additional risk factor for disease and fibrosis progression. The study aims to evaluate whether a therapy with direct-acting antiviral agents leading to a sustained virologic response directly impacts parameters reflecting glucose metabolism and fibrosis.

DETAILED DESCRIPTION:
Chronic hepatitis C infection is associated with changes of glucose metabolism end increased frequency of impaired glucose tolerance. It is well known that metabolic factors play an important role in fibrosis progression and steatohepatitis for example in non-alcoholic steatohepatitis (NASH). Accordingly changes in glucose metabolism in patients with chronic hepatitis C might directly impact disease and fibrosis progression. The study aims to evaluate whether a therapy with direct-acting antiviral agents leading to a sustained virologic response directly impacts parameters reflecting glucose metabolism and fibrosis. Follow-up examinations will determine the long-term metabolic changes of successful elimination of the virus by antiviral treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic hepatitis C infection and planned antiviral therapy with direct-acting antiviral agents
2. Age 18-99
3. Informed Consent

Exclusion Criteria:

1. Patients without legal capacity for informed consent
2. alcohol intake ≥ 20 g/d (f) und 30 g/d (m) within one year of study screening
3. Decompensated cirrhosis
4. viral co-infection
5. HIV infection
6. Non-viral chronic liver disease
7. Malignancy within 5 years before study screening except basalioma
8. liver transplant recipients
9. weight loss ≥10% within 3 months before study screening
10. Changes of diabetic drug treatment, lipid lowering therapy oder vitamin E within three months before study screening.
11. Intake of medication associated with hepatic steatosis (e.g. steroids, methotrexate, amiodarone, tamoxifen, valproat, flutamide, tetracyclins, cytostatics etc.)
12. Bariatric surgery in personal history
13. Clinically relevant congestive heart disease, cardiac arrythmia, valvular heart disease)
14. Implanted cardiac pacemaker or defibrillator
15. Patients during pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C infection with planned antiviral DAA treatment
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients with changes in glucose metabolism measured by fasting glucose | From baseline up to one year after end of treatment
  rate of patients with normal fasting glucose (<100mg/dl), prediabetes (glucose 100-125mg/d) and diabetes (>126mg/dl)
Rate of patients with changes in glucose metabolism measured by Homeostasis Model Assessment-index (HOMA) | From baseline up to one year after end of treatment
  Homeostasis Model Assessment-index (HOMA) measures insulin resistance:
  1. <2,0 insulin resistance unlikely
  2. 2,0 - 2,5 insulin resistance possible
  3. 2,5 - 5,0 insulin resitance likely
  4. >5,0 proven insulin resitance
Rate of patients with changes in glucose metabolism measured by HbA1c | From baseline up to one year after end of treatment
  rate of patients with normal HbA1c (>6% Hb), prediabetes (6-6.4% Hb) and diabetes (>6.5% Hb)

SECONDARY OUTCOMES:
Liver fibrosis 1 | From baseline up to one year after end of treatment
  Evaluation of changes of parameters reflecting liver fibrosis: Fibroscan
Liver fibrosis 2 | From baseline up to one year after end of treatment
  Evaluation of changes of parameters reflecting liver fibrosis: ARFI

CONTACTS AND LOCATIONS:
Overall Officials: Tania Welzel, MD, Principal Investigator — Prof.
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No